CLINICAL TRIAL: NCT00423124
Title: A Phase I-II Study: Infusion of Donor Lymphocytes Transduced With the Suicide Gene HSV TK, After Transplantation of Allogeneic T-depleted Stem Cells From a Haploidentical Donor in Patients With Haematological Malignancies
Brief Title: Infusion of Donor Lymphocytes Transduced With the Suicide Gene HSV TK in Patients With Haematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK007; 2005-003587-34 (EudraCT Number)
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Hematological Malignancies
Keywords: Hematological malignancies; HSV-TK; Haploidentical HCT; GvHD; GvL
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Genetic: HSV-TK

INTERVENTIONS:
Genetic: HSV-TK — Infusion of genetically modified lymphocytes (1x10^6-1x10^7 c/kg): first at +21-+49 days after HSCT; in absence of immune reconstitution and GvHD further infusions up to 4 will be administered on monthly basis.

SUMMARY:
The aim of the study is to obtain immune reconsitutuion as well as reduction of infective episodes and disease relapse in patient with haematological malignancies who underwent SCT(and subsequent T lymphocytes infusions) and selectively controlling GvHD.

DETAILED DESCRIPTION:
Delayed immune-reconstitution remains one of the main limitation of haploidentical stem cell transplantation. The risk of severe infections remains high for several months and CD4+ reconstitution could take more than 10 months. The low number of lymphocytes infused with the graft, the degree of HLA disparity, and a reduced thymic function in adults and differences in host/donor antigen presenting cells are contributing causes.

The infusions of HSV-TK engineered lymphocytes may represent a significant therapeutic improvement in haploidentical haplo-HCT, because it remarkably may enhance both GvL activity, thus reducing the occurrence of disease relapse, and post-transplant immune reconstitution in the absence of chronic immune suppression, thus decreasing the rate of both post-transplant opportunistic infections and transplant-related mortality. Furthermore, the efficient control of GvHD achieved via the suicide mechanism allows also the multiple infusion of HSV-TK-treated donor lymphocytes, when needed, that might further improve post-transplant host immune reconstitution, and, eventually, survival in patients receiving haplo-HCT. Finally, this therapeutic approach, which allows the safe infusion of escalating doses of donor lymphocytes, can become a valuable option for all candidates, including patients with advanced disease and older age.

The proposed clinical trial represents an innovative therapeutic treatment for patients affected by hematological malignancies, who have undergone haploidentical stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients >=18 years old affected by hematological malignancies at high risk of relapse based on disease progression or presence of negative prognostic factors, who have received a HCT from donor HLA mismatched (haploidentical) for 2 or 3 loci
* Engraftment documented by >500 neutrophils/µl for three consecutive days in the absence of growth factors
* Mixed chimerism or full donor chimerism confirmed
* AML in 1st or 2nd relapse or primary refractory
* High-risk AML in 1st or subsequent remission
* RAEB and RAEB-T
* CML in 2nd chronic phase, blast crisis or accelerated phase
* Poor prognosis ALL in 1st or subsequent remission
* High grade lymphomas in 3rd or subsequent remission
* Multiple myeloma in advanced stage relapsing or progressing after high dose chemotherapy
* Absence of fully HLA matched or one HLA locus mismatched family donor
* Stable clinical conditions and life expectancy >3 months
* PS Karnofsky >70
* Written donor/patient informed consent

Exclusion Criteria:

* Infection with cytomegalovirus being treated with ganciclovir
* Presence of GvHD grade > I that requires systemic immunosuppressive therapy (at baseline)
* Ongoing systemic immunosuppressive therapy
* Ongoing acyclovir administration
* Administration after haplo-HCT of G-CSF and cyclosporine A
* CD3+ lymphocytes >100/µl before day +42 after haplo-HCT
* Life-threatening condition or complication other than their basic disease
* CNS disease
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2002-07; Primary Completion 2011-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of clinical activity in terms of immune-reconstitution, provided by the add- back of the transduced T-cells after haplo-HCT | during the study
Evaluation of the "in vivo" control of GvHD after administration of ganciclovir in patients treated with HSV-TK transduced T-cells | during the study
Evaluation of GvL effect | during the study

SECONDARY OUTCOMES:
Time to relapse, time to death (evaluated by disease free survival and overall survival) | during the study
Incidence of infectious events (measured by number of infectious events) | during the study
Acute and long term toxicity related to the infusions (measured by incidence of adverse events) | during the study and study follow up

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Ciceri, MD, Principal Investigator — Hematology and BMT Unit, San Raffaele Scientific Institute, Milan, Italy
Locations (8):
- Medizinische Hoschule Hannover, Hanover, Germany
- G. Papanicolau, Thessaloniki, Greece
- Hadassah University Hospital, Jerusalem, Israel
- Italy (4):
  - Fondazione San Raffaele, Milan
  - Istituto Clinico Humanitas, Milan
  - Policlinico Monteluce, Perugia
  - Ospedale Civile, Pescara
- Hammersmith Hospital, London, United Kingdom

REFERENCES:
- [Result] Ciceri F, Bonini C, Stanghellini MT, Bondanza A, Traversari C, Salomoni M, Turchetto L, Colombi S, Bernardi M, Peccatori J, Pescarollo A, Servida P, Magnani Z, Perna SK, Valtolina V, Crippa F, Callegaro L, Spoldi E, Crocchiolo R, Fleischhauer K, Ponzoni M, Vago L, Rossini S, Santoro A, Todisco E, Apperley J, Olavarria E, Slavin S, Weissinger EM, Ganser A, Stadler M, Yannaki E, Fassas A, Anagnostopoulos A, Bregni M, Stampino CG, Bruzzi P, Bordignon C. Infusion of suicide-gene-engineered donor lymphocytes after family haploidentical haemopoietic stem-cell transplantation for leukaemia (the TK007 trial): a non-randomised phase I-II study. Lancet Oncol. 2009 May;10(5):489-500. doi: 10.1016/S1470-2045(09)70074-9. Epub 2009 Apr 1. PMID 19345145
- [Derived] Stornaiuolo A, Valentinis B, Sirini C, Scavullo C, Asperti C, Zhou D, Martinez De La Torre Y, Corna S, Casucci M, Porcellini S, Traversari C. Characterization and Functional Analysis of CD44v6.CAR T Cells Endowed with a New Low-Affinity Nerve Growth Factor Receptor-Based Spacer. Hum Gene Ther. 2021 Jul;32(13-14):744-760. doi: 10.1089/hum.2020.216. Epub 2021 May 5. PMID 33554732